CLINICAL TRIAL: NCT05090501
Title: A Randomized Trial of High Intensity Circuit Training in Nature and Indoors to Compare Exercise Performance, Emotions, Perceived Exertion, and the Variability of Movement and Heart Rate in Recreational Exercisers.
Brief Title: The Effects of High Intensity Circuit Training in Nature Vs. Indoor on Exercise Performance, and Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Henrique Brito, Researcher, Faculdade de Motricidade Humana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HICT in nature and indoor
Record Dates: First submitted 2021-09-29; First posted 2021-10-22 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Green Exercise; Indoor Exercise
Keywords: Nature-based exercise; Indoor exercise; High Intensity Circuit Training; Performance; Movement Variability; Affect; Perceived exertion; Heart Rate Variability; Arousal

STUDY DESIGN:
Intervention Model Description: This trial is designed as a randomised, controlled, participant blinded, superiority trial with two groups. Randomization will be performed as block randomization with a 1:1 allocation.
Who Masked: Participant, Care Provider
Masking Description: Participants will not be informed of the opposite group details, and it is not expected that they meet other participants during the meeting or intervention periods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green (Experimental): Green exercise participants will exercise in the nature-based condition.
  Interventions: Behavioral: High Intensity Circuit Training
- Indoor (Experimental): Indoor participants will exercise in the indoor condition.
  Interventions: Behavioral: High Intensity Circuit Training

INTERVENTIONS:
Behavioral: High Intensity Circuit Training — The participants will execute a 12-exercise High Intensity Circuit Training protocol. Each exercise will have an active part taking 30 seconds, in which exercisers are encouraged to do as many repetitions as possible, and a resting part taking 10 seconds in which the participants rest and are informed of the next exercise. Before and after the 12-exercise routine, the participants rate their affect, arousal and perceived exertion, while using a heart rate monitor and two IMU sensors on their arms and legs.

SUMMARY:
Exercising in a nature setting has been credited with benefits for health and well-being, more so than exercising indoors. Additionally, motoric performance in the same exercise (e.g., running speed, more strenuous physical activity) has been reported in some studies to be greater if practiced outdoors, in a nature setting. The explanation may be in the inherent variability of natural landscapes, the textures, elevations, obstacles and objects which are not found in standard built and indoor settings. Indoor settings are characterized by safe, organized, patterned textures and objects created for specific ends, which inhibit variability in physical and physiological behavior. Variability in the environment turns into variability in body systems, which benefits health, well-being, and skill acquisition.

Variability in behavior depends also on the task. Running or walking is essentially a journey throughout the environment in which interaction with obstacles, puddles, and other runners is part of the variability of the activity. On the other hand, physical activity such as HICT is done in a small area, and is a scripted, prescribed activity (e.g., push-ups, sit-ups), which lowers the amount of variability in behavior. The aim of this trial is to test if a low variability activity shows differences in performance, wellbeing, and behavior measures according to the amount of variability in the environment.

In this trial the participants will engage in two high intensity circuit training (HICT) interventions - one in an indoor setting, and another in a nature setting. The HICT intervention includes 12 calisthenic exercises, and will be performed at a self-selected intensity by the participants. Each exercise will be performed during one minute, followed by 30 seconds of rest where the participants will be instructed what the next exercise will be. Before exercising, the participants put a heart rate monitor and two inertial measurement units (IMUs) on the right arm and leg, according to the correct usage guidelines, and rate their positive affect, arousal, and perceived exertion. Immediately after exercising, they rate the same measures again.

Research Hypotheses:

Greater movement variability, heart rate variability, performance, wellbeing, and arousal during HICT in nature setting than indoor setting.

DETAILED DESCRIPTION:
Introduction: Nature environments are "any outdoor spaces that retain noticeable elements of nature, ranging from pristine or seminatural areas to urban green or blue spaces, including green infrastructure". Exercising in nature settings has been shown to improve well-being outcomes such as lower anxiety and greater positive mood, more so than exercising in artificial environments like urban spaces or indoors.

Over the past decades, the well-being benefits of nature-based exercise have been extensively reported in the literature, but exercise and sport performance have not been studied as much, in spite of some studies showing that performance may be better in natural settings than indoor conventional settings (e.g., dancing more vigorously, more power in cycling, ability to run more distance until exhaustion). This raises the question of how nature may impact performance efficacy (the product of performance, i.e., running faster) and efficiency (the psychological and physiological processes that may enhance performance efficacy) in exercise and sport activities, especially since many studies show, for example, that achieving the same goal in nature is less effortful than doing the same activity indoors.

The relationship between the exercise factor and the environment factor for potential health and performance benefits can be seen as sub-additive (less than total independent benefits of both exposures), additive (equal to the sum of the parts), and synergistic (greater than the sum of the parts).

Mechanisms: The mechanism by which physical activity in nature environments induces greater health and may enhance performance is not yet fully understood. Historically, the exercise and sport communities have created "proper" spaces to undertake their physical activities, such as gyms, stadiums, tracks. However, these standardized and artificial spaces are believed to offer limited variability in action. The ecological dynamics perspective views nature settings as a more varied and challenging landscape of affordances (possibilities for action) than that of built environments. Variability in the environment turns into variability in body systems, allowing for degenerate behavior (changing movement structure without compromising functionality). Assuming that the nature environment presents a richer and more variable landscape of affordances to exercisers has given birth to a theory within the ecological dynamics framework, labelled EVA, or the Empowering Variability of Affordances of Nature. To this end, EVA assumes that the uneven surfaces, objects and obstacles of nature settings such as grassland and trees allow for more variable athletic behavior, which has been deemed beneficial for exercise and sport performance. It must not be a coincidence that activities mostly practiced in natural environments such as extreme sports, are notorious for their demand for adaptability and creativity, and for promoting health.

Furthermore, for exercisers, the nature environment is known to elicit dissociative/exteroceptive attentive focus (i.e., focus on the environment), while the built/indoor environment elicits associative attentive focus (i.e., focus on the task itself). An associative cognitive process (focus on the task) is known to cause lower affective responses and greater exertion during exercise, particularly in high intensity physical activities. In short, exercising in nature may improve wellbeing and athletic performance due to inherent variability in action, and by eliciting exteroceptive attentive focus.

Need for a trial: Variability in behavior depends also on the task. Running or walking is essentially a journey throughout the environment in which interaction with obstacles, puddles, and other runners is part of the variability of the activity. However, HICT is done in a small area, and is a scripted, prescribed activity, lowering the amount of variability in behavior (e.g., push-ups, sit-ups). Thus, the aim of this study is to test if a closed circuit, scripted, anaerobic exercise (HICT) shows differences in movement variability, performance, and wellbeing, depending on the exercise environment (nature vs. indoor), in healthy, fit adults.

Familiarization session: Each participant goes individually to the Sport Expertise Laboratory (Spertlab) in Faculdade de Motricidade Humana and delivers the Informed Consent. The investigator then places the chest band (Polar H10) on the participant according to the correct usage guidelines, for familiarization purposes.

The participant is then shown and instructed on the Greenness Rating Scale and International Physical Activity Questionnaire (baseline questionnaires), followed by the Feeling Scale, Felt Arousal Scale, and Rating of Perceived Exertion (pre- and post-exercise measurement scales). Then the investigator demonstrates all the exercises planned for the exercise sessions, explaining to the participant the correct way to perform each one. The investigators remind that the participant should not exercise for 24 hours before the exercise sessions, and schedule two exercise sessions 48 hours apart (to prevent carry-over effects) in the following two weeks. Finally, the investigators collect the chest band and inform the participants that they must avoid ingesting caffeine, alcohol, and practicing high intensity physical activity in the 24 hours prior to the intervention sessions, and avoid ingesting food and liquids (except water) in the 3 hours prior to the sessions.

Placement of the Inertial Measurement Units (IMUs): Two IMUs are placed at the midpoint between the lateral epicondyle and the greater tubercle of the humerus, and between the lateral epicondyle and the greater trochanter of the femur, both on the right side. The upper (UL) and lower limbs (LL) are the body segments with greater activity during these calisthenic exercises; additionally, the proximal segment of the limbs is biarticular and does not run the risk of being fixed to the ground, as is the case of the hands/forearms during push-ups, and the feet/legs during squats, which would reduce the range of motion, and consequently have lesser detectable acceleration.

Intervention: As the exercise session approaches, the investigators get in touch to remind the participants about the session, to bring comfortable clothes (sports equipment). On the appointed day and time, the investigators and the participants meet at Faculdade de Motricidade Humana (FMH), and are escorted to the exercise site (Spertlab if indoor, Jamor park if outdoor). The investigators place the IMUs and the chest band on the participants as defined, deliver the Greenness Rating Scale, Feeling Scale, Felt Arousal Scale, and Rating of Perceived Exertion (available on a tablet or paper support) and inform participants that they can exercise at whatever pace they wish. The exercise session is made of 12 calisthenic exercises and is 20 minutes long (60 seconds active and 30 seconds resting per exercise), including warm-up and cool-down. The exercise session intervention will be conducted by a certified fitness instructor who will not know the objectives of the study (blinding). Exercise times will be controlled by the instructor, who will remind and if needed demonstrate to the participants what the next exercise is during the rest periods. Immediately after performing the exercises, before cool-down, participants complete the Rating of Perceived Exertion, and after returning to calm, they complete the remaining post-exercise questionnaires, and the investigators collect the chest bands and IMUs. After the session, the investigators accompany the participants again to FMH, confirm the next session in a minimum of 48 hours, and answer any queries. Participants who performed the indoor session will do the next session outdoors, and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Fit for engaging in intense physical activity according to a physician.

Exclusion Criteria:

* Participating in another research project at the same time.
* Unable to perform the proposed exercises due to physical impairment.
* Taking medication or being under medical treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | through study completion, an average of 10 minutes
  Heart Rate Variability is the variation in R-R intervals (time between systolic injections) of the heart. Heart bands will be used to collect the base R-R intervals
Movement Variability | through study completion, an average of 10 minutes
  changes in acceleration of body segments can be seen as a direct measure of body movement adaptation to environmental constraints.

SECONDARY OUTCOMES:
Exercise performance | through study completion, an average of 10 minutes
  All exercises in the intervention have cyclical concentric and eccentric phases, which will be apparent in the IMU (gyroscope) time-series. When angular velocity in any axis (x,y,z) becomes zero, and direction changes in the opposite way, it is possible to count repetitions in the specific exercise. Alternatively, the investigators will count and register the number of repetitions by notation. The final value per exercise will be a measure of the performance of the individual in that specific exercise.
Change score of the Feeling Scale | through study completion, an average of 10 minutes
  Feeling Scale (FS): Affective responses to exercise will be collected with the Feeling Scale (Hardy & Rejeski, 1989). The scale allows the measurement of mood fluctuations during exercise through a single item "How are you feeling now", in which subjects respond on a scale from -5 ("very bad") to +5 "very good", 0 being "neutral". The scale shows high reliability and validity (Emanuel et al., 2021).The scale was built to assess affective states during exercise and has been widely used in comparative studies of exercise environments.
Change score of the Rating of Perceived Exertion | through study completion, an average of 10 minutes
  Rating of Perceived Exertion (RPE): This scale is extensively used in exercise and sport research. It is a scale ranging from 6 (no exertion) to 20 (maximum exertion).
Change Score in the Trail Making Test | through study completion, an average of 10 minutes
  The Trail Making Test is a state-test of cognitive attention.

CONTACTS AND LOCATIONS:
Overall Officials: Henrique Brito, MSc, Principal Investigator — Faculdade de Motricidade Humana
Locations (1):
- Faculdade de Motricidade Humana, Cruz Quebrada, Oeiras, Portugal

IPD SHARING:
Plan to Share IPD: Yes
plan available at https://www.sciencedirect.com/science/article/pii/S1469029224000372
Supporting Information: Analytic Code
Time Frame: Data available indefinitely.
Access Criteria: Open access
URL: https://data.mendeley.com/datasets/6rfnsxsn8h/2

REFERENCES:
- [Background] Lahart I, Darcy P, Gidlow C, Calogiuri G. The Effects of Green Exercise on Physical and Mental Wellbeing: A Systematic Review. Int J Environ Res Public Health. 2019 Apr 15;16(8):1352. doi: 10.3390/ijerph16081352. PMID 30991724
- [Background] Thompson Coon J, Boddy K, Stein K, Whear R, Barton J, Depledge MH. Does participating in physical activity in outdoor natural environments have a greater effect on physical and mental wellbeing than physical activity indoors? A systematic review. Environ Sci Technol. 2011 Mar 1;45(5):1761-72. doi: 10.1021/es102947t. Epub 2011 Feb 3. PMID 21291246
- [Background] Bowler DE, Buyung-Ali LM, Knight TM, Pullin AS. A systematic review of evidence for the added benefits to health of exposure to natural environments. BMC Public Health. 2010 Aug 4;10:456. doi: 10.1186/1471-2458-10-456. PMID 20684754
- [Background] Byrka, K., & Ryczko, N. (2018). Positive effects of dancing in natural versus indoor settings: The mediating role of engagement in physical activity. Journal of Environmental Psychology, 57, 25-33. https://doi.org/10.1016/j.jenvp.2018.06.002
- [Background] Rogerson M, Barton J. Effects of the Visual Exercise Environments on Cognitive Directed Attention, Energy Expenditure and Perceived Exertion. Int J Environ Res Public Health. 2015 Jun 30;12(7):7321-36. doi: 10.3390/ijerph120707321. PMID 26133125
- [Background] Slapsinskaite, A., Garcia, S., Razon, S., Balague, N., Hristovski, R., & Tenenbaum, G. (2016). Cycling outdoors facilitates external thoughts and endurance. Psychology of Sport and Exercise, 27, 78-84. https://doi.org/10.1016/j.psychsport.2016.08.002
- [Background] Araújo, D., Brymer, E., Brito, H., Withagen, R., & Davids, K. (2019). The empowering variability of affordances of nature: Why do exercisers feel better after performing the same exercise in natural environments than in indoor environments? Psychology of Sport and Exercise, 42, 138-145. https://doi.org/10.1016/j.psychsport.2018.12.020
- [Background] Exel J, Mateus N, Goncalves B, Abrantes C, Calleja-Gonzalez J, Sampaio J. Entropy Measures Can Add Novel Information to Reveal How Runners' Heart Rate and Speed Are Regulated by Different Environments. Front Psychol. 2019 Jun 4;10:1278. doi: 10.3389/fpsyg.2019.01278. eCollection 2019. PMID 31214084
- [Background] Moras G, Fernandez-Valdes B, Vazquez-Guerrero J, Tous-Fajardo J, Exel J, Sampaio J. Entropy measures detect increased movement variability in resistance training when elite rugby players use the ball. J Sci Med Sport. 2018 Dec;21(12):1286-1292. doi: 10.1016/j.jsams.2018.05.007. Epub 2018 May 24. PMID 29804653
- [Background] Klika, B., & Jordan, C. (2013). High-intensity circuit training using body weight: maximum Results With Minimal Investment. ACSM's Health & Fitness Journal, 17(3), 8-13. https://doi.org/10.1249/FIT.0b013e31828cb1e8
- [Background] Silva RA, Rogers K, Buckley TJ. Advancing Environmental Epidemiology to Assess the Beneficial Influence of the Natural Environment on Human Health and Well-Being. Environ Sci Technol. 2018 Sep 4;52(17):9545-9555. doi: 10.1021/acs.est.8b01781. Epub 2018 Aug 24. PMID 30064205
- [Background] Flowers, E. P., Freeman, P., & Gladwell, V. F. (2018). Enhancing the acute psychological benefits of green exercise: An investigation of expectancy effects. Psychology of Sport and Exercise, 39, 213-221. https://doi.org/10.1016/j.psychsport.2018.08.014
- [Background] Jang, S., & So, W.-Y. (2017). The effect of short-term outdoor taekwondo training on the concentration and mood of taekwondo players. Journal of Men's Health, 13(2), e68-e75. https://doi.org/10.22374/1875-6859.13.2.9
- [Background] Niedermeier M, Grafetstatter C, Hartl A, Kopp M. A Randomized Crossover Trial on Acute Stress-Related Physiological Responses to Mountain Hiking. Int J Environ Res Public Health. 2017 Aug 11;14(8):905. doi: 10.3390/ijerph14080905. PMID 28800067
- [Background] Shanahan DF, Franco L, Lin BB, Gaston KJ, Fuller RA. The Benefits of Natural Environments for Physical Activity. Sports Med. 2016 Jul;46(7):989-95. doi: 10.1007/s40279-016-0502-4. PMID 26886475
- [Background] Brymer E, Araujo D, Davids K, Pepping GJ. Conceptualizing the Human Health Outcomes of Acting in Natural Environments: An Ecological Perspective. Front Psychol. 2020 Jul 16;11:1362. doi: 10.3389/fpsyg.2020.01362. eCollection 2020. PMID 32765336
- [Background] Donnelly AA, MacIntyre TE, O'Sullivan N, Warrington G, Harrison AJ, Igou ER, Jones M, Gidlow C, Brick N, Lahart I, Cloak R, Lane AM. Environmental Influences on Elite Sport Athletes Well Being: From Gold, Silver, and Bronze to Blue Green and Gold. Front Psychol. 2016 Aug 4;7:1167. doi: 10.3389/fpsyg.2016.01167. eCollection 2016. PMID 27540370
- [Background] Collins, L., & Brymer, E. (2020). Understanding nature sports: a participant centred perspective and its implications for the design and facilitating of learning and performance. Annals of Leisure Research, 23(1), 110-125. https://doi.org/10.1080/11745398.2018.1525302
- [Background] Reich AH, Queathem EJ. Setting, Age, and Intensity Influence Responses to Exercise in Young Endurance Runners. Percept Mot Skills. 2020 Jun;127(3):533-554. doi: 10.1177/0031512520903907. Epub 2020 Feb 9. No abstract available. PMID 32036749
- [Background] Hutchinson, J. C., & Tenenbaum, G. (2007). Attention focus during physical effort: The mediating role of task intensity. Psychology of Sport and Exercise, 8(2), 233-245. https://doi.org/https://doi.org/10.1016/j.psychsport.2006.03.006
- [Background] Lind E, Welch AS, Ekkekakis P. Do 'mind over muscle' strategies work? Examining the effects of attentional association and dissociation on exertional, affective and physiological responses to exercise. Sports Med. 2009;39(9):743-64. doi: 10.2165/11315120-000000000-00000. PMID 19691364
- [Derived] Brito H, Lopes H, Vaz de Carvalho M, Carrilho D, Carvalho A, Araujo D. The effects of nature-based vs. indoor settings on the adaptability, performance and affect of calisthenics exercisers. A registered report. Psychol Sport Exerc. 2024 Jul;73:102626. doi: 10.1016/j.psychsport.2024.102626. Epub 2024 Mar 15. PMID 38492765